CLINICAL TRIAL: NCT00336323
Title: A Phase 2 Evaluation of Anti-VEGF Therapy for Diabetic Macular Edema: Bevacizumab (Avastin)
Acronym: Bevacizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Roy W. Beck, M.D., Ph.D., Director, Jaeb Center for Health Research (DRCR.net)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEI-129; U10EY018817-03 (NIH); U10EY014229-07 (NIH); U10EY014231-09 (NIH); EY14231, EY14269, EY14229
Record Dates: First submitted 2006-06-09; First posted 2006-06-13 (Estimated); Results first posted 2011-07-12 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic; macular; edema; avastin; bevacizumab; anti-VEGF; retinal thickness; visual acuity; DME
MeSH Terms: conditions — Diabetic Retinopathy; Edema | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Active Comparator): Laser photocoagulation at baseline
  Interventions: Procedure: Laser Photocoagulation
- 2 (Experimental): 1.25 mg intravitreal injection of bevacizumab at baseline and 6 weeks
  Interventions: Drug: Bevacizumab
- 3 (Experimental): 2.5 mg intravitreal injection of bevacizumab at baseline and 6 weeks
  Interventions: Drug: Bevacizumab
- 4 (Experimental): 1.25 mg intravitreal injection of bevacizumab at baseline (sham injection at 6 weeks)
  Interventions: Drug: Bevacizumab
- 5 (Experimental): 1.25 mg intravitreal injection of bevacizumab at baseline, laser photocoagulation at 3 weeks, and intravitreal injection of 1.25 mg bevacizumab at 6 weeks
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Procedure: Laser Photocoagulation — Laser photocoagulation at baseline; If edema present at 12 weeks, can be treated with 2 intravitreal injections of 1.25 mg bevacizumab spaced 6 weeks apart
  Arms: 1
Drug: Bevacizumab — 1.25 mg intravitreal injection of bevacizumab at baseline and 6 weeks
  Other Names: Avastin; anti-VEGF drug
  Arms: 2
Drug: Bevacizumab — 2.5 mg intravitreal injection of bevacizumab at baseline and 6 weeks
  Other Names: Avastin; anti-VEGF drug
  Arms: 3
Drug: Bevacizumab — 1.25 mg intravitreal injection of bevacizumab at baseline (sham injection at 6 weeks)
  Other Names: Avastin; anti-VEGF drug
  Arms: 4
Drug: Bevacizumab — 1.25 mg intravitreal injection of bevacizumab at baseline, laser photocoagulation at 3 weeks, and intravitreal injection of 1.25 mg bevacizumab at 6 weeks
  Other Names: Avastin; anti-VEGF drug
  Arms: 5

SUMMARY:
This study will provide preliminary data on the dose and dose interval related effects of intravitreally administered Avastin on retinal thickness and visual acuity in subjects with Diabetic Macular Edema (DME) to aid in planning a phase 3 trial.

In addition, this study will provide preliminary data on the safety of intravitreally administered Avastin in subjects with DME.

DETAILED DESCRIPTION:
Diabetic retinopathy is a major cause of visual impairment in the United States. Diabetic macular edema (DME) is a manifestation of diabetic retinopathy that produces loss of central vision. Data from the Wisconsin Epidemiologic Study of Diabetic Retinopathy (WESDR) estimate that after 15 years of known diabetes, the prevalence of diabetic macular edema is approximately 20% in patients with type 1 diabetes mellitus (DM), 25% in patients with type 2 DM who are taking insulin, and 14% in patients with type 2 DM who do not take insulin.

In a review of three early studies concerning the natural history of diabetic macular edema, Ferris and Patz found that 53% of 135 eyes with diabetic macular edema, presumably all involving the center of the macula, lost two or more lines of visual acuity over a two year period. In the Early Treatment Diabetic Retinopathy Study (ETDRS), 33% of 221 untreated eyes available for follow-up at the 3-year visit, all with edema involving the center of the macula at baseline, had experienced a 15 or more letter decrease in visual acuity score (equivalent to a doubling of the visual angle, e.g., 20/25 to 20/50, and termed "moderate visual loss").

In the ETDRS, focal photocoagulation (direct treatment to microaneurysms and grid treatment to diffuse edema) of eyes with clinically significant macular edema (CSME) reduced the risk of moderate visual loss by approximately 50% (from 24% to 12%, three years after initiation of treatment). Therefore, 12% of treated eyes developed moderate visual loss in spite of treatment. Furthermore, approximately 40% of treated eyes that had retinal thickening involving the center of the macula at baseline still had thickening involving the center at 12 months, as did 25% of treated eyes at 36 months.

Although several treatment modalities are currently under investigation, the only demonstrated means to reduce the risk of vision loss from diabetic macular edema are laser photocoagulation, as demonstrated by the ETDRS, intensive glycemic control, as demonstrated by the Diabetes Control and Complications Trial (DCCT) and the United Kingdom Prospective Diabetes Study (UKPDS) and blood pressure control, as demonstrated by the UKPDS. In the DCCT, intensive glucose control reduced the risk of onset of diabetic macular edema by 23% compared with conventional treatment. Long-term follow-up of patients in the DCCT show a sustained effect of intensive glucose control, with a 58% risk reduction in the development of diabetic macular edema for the DCCT patients followed in the Epidemiology of Diabetes Interventions and Complications Study.

The frequency of an unsatisfactory outcome with respect to proportion with vision improvement following laser photocoagulation in some eyes with diabetic macular edema has prompted interest in other treatment modalities. One such treatment is pars plana vitrectomy. These studies suggest that vitreomacular traction, or the vitreous itself, may play a role in increased retinal vascular permeability. Removal of the vitreous or relief of mechanical traction with vitrectomy and membrane stripping may be followed by substantial resolution of macular edema and corresponding improvement in visual acuity. However, this treatment may be applicable only to a specific subset of eyes with diabetic macular edema that have a component of vitreomacular traction contributing to the edema. It also requires a complex surgical intervention with its inherent risks, recovery time, and expense. Other treatment modalities such as pharmacologic therapy with oral protein kinase C inhibitors and use of intravitreal corticosteroids are under investigation. The use of antibodies targeted at vascular endothelial growth factor (VEGF), such as in the current study, is another treatment modality that has generated considerable interest, and is currently being investigated in phase 3 trials of choroidal neovascularization in age-related macular degeneration (with pegaptanib or ranibizumab) or diabetic macular edema (with pegaptanib).

Increased VEGF levels have been demonstrated in the retina and vitreous of human eyes with diabetic retinopathy. VEGF, also known as vascular permeability factor, has been demonstrated to increase vessel permeability by increasing the phosphorylation of tight junction proteins, and has been shown to increase retinal vascular permeability in in vivo models. Anti-VEGF therapy, therefore, may represent a useful therapeutic modality which targets the underlying pathogenesis of diabetic macular edema.

Bevacizumab is currently approved for the treatment of metastatic colorectal cancer, and published case reports and widespread clinical use have suggested its efficacy in the treatment of neovascular age-related macular degeneration and macular edema associated with diabetes and central retinal vein occlusion. To date, no evidence of ocular inflammation or other adverse events has been noted in association with intravitreal injection of bevacizumab. However, a study has not been conducted to evaluate its efficacy and safety. In view of the widespread use of bevacizumab, such a study is important to conduct.

From a public health perspective, an intravitreal bevacizumab study is also important to conduct because of the relatively low cost of the bevacizumab drug. As noted earlier, bevacizumab is marketed for systemic use for colon cancer. The dose used in the eye is a fraction of the systemic dose and costs $25 to $50 per dose.

The two doses of bevacizumab being evaluated in this study will be 1.25 mg, which is the dose that has most commonly been used in clinical practice, and 2.5 mg, which has also been used though less commonly. A lower dose than 1.25 mg would create difficulties with dilution and the accuracy of injection of a small volume.

The optimal interval for the bevacizumab doses is not known. Six weeks has been selected for this study as it is not believed that the effect will last longer than this. Retinal thickening and visual acuity will be measured at 3 and 6 weeks to provide the requisite information to judge the duration of effect.

There is expected to be a beneficial cumulative effect of multiple doses. A total of two doses, spaced 6 weeks apart, was selected for the study with the primary outcome 3 weeks after the second dose.

The decision as to whether to proceed to a phase 3 trial will be based on the observation of a substantial reduction in retinal thickening in the bevacizumab-treated eyes compared with the laser-treated eyes and at least a suggestion of benefit on visual acuity, plus a safety profile of minimal risk.

Description: The study involves the enrollment of subjects over 18 years of age with diabetic macular edema. Subjects will have one study eye randomly assigned with equal probability (stratified by visual acuity) to one of 5 treatment groups:

Laser photocoagulation at baseline

1.25 mg intravitreal injection of bevacizumab at baseline and 6 weeks

2.5 mg intravitreal injection of bevacizumab at baseline and 6 weeks

1.25 mg intravitreal injection of bevacizumab at baseline (sham injection at 6 weeks)

1.25 mg intravitreal injection of bevacizumab at baseline, laser photocoagulation at 3 weeks, and intravitreal injection of 1.25 mg bevacizumab at 6 weeks

Follow-up includes 10 visits at 4 days, 3 weeks, 6 weeks, 4 days following 6 weeks, 9 weeks, 12 weeks, 18 weeks, 24 weeks, 41 weeks and 70 weeks. At each visit, visual acuity and ocular exams are completed on both eyes, and an OCT is performed on the study eye (except at the 4-day visits).

During the first 12 weeks, no other treatment for DME is given. During weeks 13-24, treatment depends on the response to the treatment given during the first 12 weeks. After 24 weeks, follow-up is for safety and treatment is at the investigator's discretion.

ELIGIBILITY:
SUBJECT-LEVEL INCLUSION CRITERIA

To be eligible, the following inclusion criteria (1-3) must be met:

1. Age >= 18 years
2. Diagnosis of diabetes mellitus (type 1 or type 2)
3. Able and willing to provide informed consent.

   EXCLUSION

   A subject is not eligible if any of the following exclusion criteria (4-13) are present:
4. Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
5. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
6. Participation in an investigational trial within 30 days of randomization that involved treatment with any drug that has not received regulatory approval at the time of study entry.
7. Known allergy to any component of the study drug.
8. Blood pressure > 180/110 (systolic above 180 OR diastolic above 110).
9. Major surgery within 28 days prior to randomization or major surgery planned during the next 6 months.
10. Myocardial infarction, other cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 6 months prior to randomization.
11. Systemic anti-VEGF or pro-VEGF treatment within 3 months prior to randomization.
12. For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 6 months.
13. Subject is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the first 6 months of the study.

STUDY EYE CRITERIA

The subject must have one eye meeting all of the inclusion criteria (a-e) and none of the exclusion criteria (f-r) listed below.

Subjects can have only one study eye. If both eyes are eligible, the study eye will be selected by the investigator and subject.

The eligibility criteria for a study eye are as follows:

INCLUSION

1. Best corrected E-ETDRS visual acuity letter score of >= 24 (i.e., 20/320 or better) and <= 78 (i.e., 20/32 or worse) within 8 days of randomization.
2. On clinical exam, definite retinal thickening due to diabetic macular edema involving the center of the macula.
3. OCT central subfield >=275 microns within 8 days of randomization.
4. Media clarity, pupillary dilation, and subject cooperation sufficient for adequate fundus photographs.
5. If prior macular photocoagulation has been performed, the investigator believes that the study eye may possibly benefit from additional photocoagulation.

   EXCLUSION

   The following exclusions apply to the study eye only (i.e., they may be present for the nonstudy eye):
6. Macular edema is considered to be due to a cause other than diabetic macular edema.
7. An ocular condition is present such that, in the opinion of the investigator, visual acuity would not improve from resolution of macular edema (e.g., foveal atrophy, pigmentary changes, dense subfoveal hard exudates, nonretinal condition).
8. An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, etc.).
9. Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal).
10. History of treatment for DME at any time in the past 3 months (such as focal/grid macular photocoagulation, intravitreal or peribulbar corticosteroids, anti-VEGF drugs, or any other treatment).
11. History of panretinal scatter photocoagulation (PRP) within 4 months prior to randomization.
12. Anticipated need for PRP in the 6 months following randomization.
13. History of prior pars plana vitrectomy.
14. History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 6 months or anticipated within the next 6 months following randomization.
15. History of YAG capsulotomy performed within 2 months prior to randomization.
16. Aphakia.
17. Uncontrolled glaucoma (in investigator's judgment).
18. Exam evidence of external ocular infection, including conjunctivitis, chalazion, or significant blepharitis.

FELLOW EYE CRITERIA

The fellow eye must meet the following criteria:

1. Best corrected E-ETDRS visual acuity letter score >= 19 (i.e., 20/400 or better).
2. No anti-VEGF treatment within the past 3 months and no expectation of such treatment in next 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2006-06; Primary Completion 2006-11 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid U. Scott, M.D., M.P.H., Study Chair — Penn State College of Medicine
Locations (34):
- United States (34):
  - Loma Linda University Health Care, Dept. of Ophthalmology, Loma Linda, California
  - Southern California Desert Retina Consultants, MC, Palm Springs, California
  - California Retina Consultants, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Retina Vitreous Consultants, Fort Lauderdale, Florida
  - Central Florida Retina Institute, Lakeland, Florida
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Illinois Retina Associates, Joliet, Illinois
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - American Eye Institute, New Albany, Indiana
  - Retina and Vitreous Associates of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Maine Vitreoretinal Consultants, Bangor, Maine
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Retina Consultants of Delmarva, P.A., Salisbury, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Retina Center, PA, Minneapolis, Minnesota
  - Charlotte Eye, Ear, Nose and Throat Assoc., PA, Charlotte, North Carolina
  - Wake Forest University Eye Center, Winston-Salem, North Carolina
  - Retina Associates of Cleveland, Inc., Beachwood, Ohio
  - Retina Northwest, PC, Portland, Oregon
  - Casey Eye Institute, Portland, Oregon
  - Penn State College of Medicine, Hershey, Pennsylvania
  - Retina Consultants, Providence, Rhode Island
  - Palmetto Retina Center, Columbia, South Carolina
  - Carolina Retina Center, Columbia, South Carolina
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - West Texas Retina Consultants P.A., Abilene, Texas
  - Retina Research Center, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Charles A. Garcia, PA & Associates, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Result] Diabetic Retinopathy Clinical Research Network; Scott IU, Edwards AR, Beck RW, Bressler NM, Chan CK, Elman MJ, Friedman SM, Greven CM, Maturi RK, Pieramici DJ, Shami M, Singerman LJ, Stockdale CR. A phase II randomized clinical trial of intravitreal bevacizumab for diabetic macular edema. Ophthalmology. 2007 Oct;114(10):1860-7. doi: 10.1016/j.ophtha.2007.05.062. Epub 2007 Aug 15. PMID 17698196
- [Result] Scott IU, Bressler NM, Bressler SB, Browning DJ, Chan CK, Danis RP, Davis MD, Kollman C, Qin H; Diabetic Retinopathy Clinical Research Network Study Group. Agreement between clinician and reading center gradings of diabetic retinopathy severity level at baseline in a phase 2 study of intravitreal bevacizumab for diabetic macular edema. Retina. 2008 Jan;28(1):36-40. doi: 10.1097/IAE.0b013e31815e9385. PMID 18185135
- [Derived] Bhavsar AR, Ip MS, Glassman AR; DRCRnet and the SCORE Study Groups. The risk of endophthalmitis following intravitreal triamcinolone injection in the DRCRnet and SCORE clinical trials. Am J Ophthalmol. 2007 Sep;144(3):454-6. doi: 10.1016/j.ajo.2007.04.011. PMID 17765429

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-six clinical sites across the United States recruited 121 subjects (109 met criteria for inclusion in the analyses) between June 2006 and August 2006.
Pre-assignment Details: Unless otherwise noted, differences in number of Participants at different visits reflect a missed visit, not a drop-out.
Groups:
- Laser at Baseline: Laser photocoagulation at baseline: If edema is present at 12 weeks, can be treated with 2 intravitreal injections of 1.25 mg bevacizumab spaced 6 weeks apart
- 1.25 mg Injection at Baseline and at 6 Weeks: 1.25 mg intravitreal injection of bevacizumab at baseline and 6 weeks
- 2.5 mg Injection at Baseline and 6 Weeks: 2.5 mg intravitreal injection of bevacizumab at baseline and 6 weeks
- 1.25 mg Injection at Baseline Only: 1.25 mg intravitreal injection of bevacizumab at baseline (sham injection at 6 weeks)
- 1.25 mg Injection at Baseline, Laser at 3w + 1.25 mg Inj at 3w: 1.25 mg intravitreal injection of bevacizumab at baseline, laser photocoagulation at 3 weeks, and intravitreal injection of 1.25 mg bevacizumab at 6 weeks
Period: Overall Study
Arm/Group | Laser at Baseline | 1.25 mg Injection at Baseline and at 6 Weeks | 2.5 mg Injection at Baseline and 6 Weeks | 1.25 mg Injection at Baseline Only | 1.25 mg Injection at Baseline, Laser at 3w + 1.25 mg Inj at 3w
Started | 19 | 22 | 24 | 22 | 22
3 Week Visit | 18 | 21 | 24 | 22 | 20 (Laser given late at six weeks for one patient)
6 Week Visit | 18 | 22 | 24 | 22 | 20 (1 patient was dropped - injection was given late at 9 wks for one patient)
9 Week Visit | 18 | 21 | 23 | 21 | 19
12 Week Visit | 19 | 21 | 24 | 22 | 20 (1 patient was dropped from study)
18 Week Visit | 19 | 22 | 23 | 21 | 18 (1 patient was dropped from the study)
24 Week Visit | 18 | 20 (1 patient was dropped from the study) | 22 (1 patient was dropped from the study) | 22 | 19
Completed | 19 | 21 | 23 | 22 | 19
Not Completed | 0 | 1 | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laser at Baseline | 1.25 mg Injection at Baseline and at 6 Weeks | 2.5 mg Injection at Baseline and 6 Weeks | 1.25 mg Injection at Baseline Only | 1.25 mg Injection at Baseline, Laser at 3w + 1.25 mg Inj at 3w | Total
Number analyzed (Participants) | 19 | 22 | 24 | 22 | 22 | 109
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [57 to 72] | 63 [54 to 73] | 68 [59 to 75] | 60 [54 to 75] | 67 [60 to 71] | 65 [57 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 9 | 9 | 10 | 43
  Male | 10 | 16 | 15 | 13 | 12 | 66
Race/Ethnicity, Customized [Number; unit: participants]
  White | 10 | 16 | 20 | 18 | 19 | 83
  African-American | 7 | 3 | 2 | 3 | 2 | 17
  Hispanic or Latino | 2 | 2 | 2 | 0 | 1 | 7
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Unknown/ not reported | 0 | 1 | 0 | 0 | 0 | 1
Character of Diabetic Macular Edema (DME) [Number; unit: participants] — Criteria used to define categories was based on investigator discretion.
  participants
    Typical/Predominantly Focal | 6 | 5 | 2 | 3 | 4 | 20
    Neither Predominantly Focal or Diffuse | 4 | 5 | 5 | 6 | 6 | 26
    Typical/Predominantly Diffuse | 9 | 12 | 17 | 13 | 12 | 63
Cystoid Abnormalities on Optical Coherence Tomography (OCT) [Number; unit: participants]
  Yes | 18 | 22 | 24 | 21 | 21 | 106
  No | 1 | 0 | 0 | 1 | 1 | 3
Diabetes Type [Number; unit: participants]
  Type 1 | 1 | 1 | 3 | 2 | 1 | 8
  Type 2 | 18 | 21 | 21 | 20 | 21 | 101
Lens status (clinical examination) [Number; unit: participants]
  Phakic | 12 | 15 | 14 | 12 | 13 | 66
  Pseudophakic | 7 | 7 | 10 | 10 | 9 | 43
Prior Panretinal Scatter Photocoagulation [Number; unit: participants]
  Yes | 3 | 2 | 3 | 1 | 4 | 13
  No | 16 | 20 | 21 | 21 | 18 | 96
Prior Treatment for Diabetic Macular Edema (DME) in Study Eye [Number; unit: participants]
  None | 7 | 5 | 10 | 5 | 7 | 34
  Focal photocoagulation alone | 4 | 11 | 9 | 6 | 9 | 39
  Focal photocoagulation plus other treatment | 8 | 3 | 3 | 11 | 6 | 31
  Other treatment without focal photocoagulation | 0 | 3 | 2 | 0 | 0 | 5
Retinopathy Severity [Number; unit: participants] — Early Treatment Diabetic Retinopathy Study Severity Scale
  participants
    Mild nonproliferative diabetic retinopathy (NPDR) | 1 | 6 | 3 | 0 | 4 | 14
    Moderate NPDR | 5 | 3 | 1 | 3 | 3 | 15
    Moderately severe NPDR | 5 | 6 | 8 | 8 | 9 | 36
    Severe NPDR | 0 | 1 | 2 | 4 | 1 | 8
    Mild proliferative diabetic retinopathy (PDR) | 4 | 5 | 6 | 5 | 4 | 24
    Moderate PDR | 1 | 0 | 2 | 0 | 1 | 4
    High Risk PDR | 2 | 0 | 0 | 0 | 0 | 2
    Missing | 1 | 1 | 2 | 2 | 0 | 6
Subretinal Fluid on Optical Coherence Tomography (OCT) [Number; unit: participants]
  Definite, center | 2 | 2 | 7 | 2 | 4 | 17
  Definite, not center | 0 | 1 | 1 | 0 | 1 | 3
  Questionable | 0 | 1 | 0 | 2 | 0 | 3
  No evidence | 16 | 18 | 16 | 18 | 17 | 85
  Missing | 1 | 0 | 0 | 0 | 0 | 1
Baseline Visual Acuity [Median (Inter-Quartile Range); unit: letter score] — Best corrected visual acuity letter score as measured by a certified tester using an electronic visual acuity testing machine based on the Early Treatment Diabetic Retinopathy Study (ETDRS) method. Best value on the scale 97, worst 0.
  letter score | 64 [50 to 70] | 65 [60 to 70] | 63 [57 to 71] | 64 [52 to 68] | 66 [57 to 72] | 64 [56 to 71]
Duaration of Diabetes [Median (Inter-Quartile Range); unit: years] | 17 [13 to 22] | 15 [8 to 22] | 18 [12 to 22] | 17 [11 to 25] | 20 [7 to 30] | 17 [11 to 23]
Hemoglobin A1c [Median (Inter-Quartile Range); unit: percent HbA1c] — Missing for 8 patients
  percent HbA1c | 7.0 [6.5 to 8.2] | 7.4 [5.9 to 7.8] | 7.3 [6.4 to 8.4] | 6.7 [6.3 to 7.4] | 7.1 [6.2 to 7.7] | 6.9 [6.3 to 8.1]
Optical Coherence Tomography (OCT) Central Subfield Thickness [Median (Inter-Quartile Range); unit: microns] | 441 [354 to 512] | 397 [320 to 538] | 446 [342 to 543] | 406 [353 to 520] | 389 [308 to 452] | 411 [334 to 505]
Optical Coherence Tomography Retinal Volume [Median (Inter-Quartile Range); unit: mm^3] | 8.3 [7.3 to 10.2] | 9.5 [8.0 to 10.3] | 9.1 [8.0 to 10.0] | 8.9 [7.7 to 10.0] | 8.6 [7.7 to 9.2] | 8.6 [7.8 to 10.1]

OUTCOME MEASURES:

1. Primary Outcome: Change in Central Subfield Retinal Thickness From Baseline Over All Study Visits
Description: Change in central subfield retinal thickness from baseline measured on Optical Coherence Tomography (OCT). OCT images were obtained at each visit following pupil dilation by a certified operator using the OCT3 machine (Carl Zeiss Meditec Inc., Dublin, CA). Scans were 6 mm length and included the 6 radial line pattern for quantitative measures and the cross hair pattern (6-12 to 9-3 o'clock) for qualitative assessment of retinal morphology. The OCT scans were sent to the DRCR.net Reading Center for grading. Negative changes represent a decrease in retinal thickening.
Time Frame: Baseline to 3,6,9, and 12 weeks
Population: The primary analysis included per protocol and intent to treat analysis. The intent to treat analysis included all randomized eyes. The last observation carried forward method was used to impute missing data. The per-protocol analysis was performed including only patients who receive treatment as per the protocol and complete the 9-week exam.
Measure: Median (Inter-Quartile Range); unit: microns
Arm/Group | Laser at Baseline | 1.25 mg Injection at Baseline and at 6 Weeks | 2.5 mg Injection at Baseline and 6 Weeks | 1.25 mg Injection at Baseline Only | 1.25 mg Injection at Baseline, Laser at 3w + 1.25 mg Inj at 3w
Number analyzed (Participants) | 19 | 22 | 24 | 22 | 22
microns
  3 Weeks | 21 [-62 to 79] | -35 [-155 to 6] | -86 [-131 to -11] | -3 [-49 to 7] | -13 [-104 to 26]
  6 Weeks | -40 [-105 to 73] | -35 [-112 to 6] | -42 [-127 to -10] | -17 [-58 to 25] | -20 [-73 to 35]
  9 Weeks | -53 [-115 to 53] | -74 [-113 to -31] | -56 [-127 to -20] | 5 [-34 to 53] | -48 [-128 to 33]
  12 Weeks | -40 [-146 to 86] | -56 [-120 to -6] | -47 [-125 to -16] | -5 [-41 to 53] | -40 [-103 to 33]
Statistical Analysis 1: Comparison: Laser at Baseline vs 1.25 mg Injection at Baseline and at 6 Weeks; Comparison of central subfield thickness at the 3 week visit between the laser only treatment group to the 1.25 mg injection at baseline and at 6 weeks treatment group; Test type: Superiority or Other; p = 0.009, Least squares regression; Adjusted for baseline values
Statistical Analysis 2: Comparison: Laser at Baseline vs 2.5 mg Injection at Baseline and 6 Weeks; Comparison of central subfield thickness at the 3 week visit between the laser only treatment group to the 2.5mg injection at baseline and 6 weeks treatment group; Test type: Superiority or Other; p < 0.001, Least squares regression; Adjusted for baseline values
Statistical Analysis 3: Comparison: 1.25 mg Injection at Baseline and at 6 Weeks vs 2.5 mg Injection at Baseline and 6 Weeks; Comparison of the reduction in central subfield thickening in the 1.25mg injection at baseline and at 6 weeks treatment group with the 2.5mg injection at baseline and 6 weeks treatment group at the 3 week visit; Test type: Superiority or Other; p = 0.66, Least squares regression — Adjusted for baseline values
Statistical Analysis 4: Comparison: 1.25 mg Injection at Baseline and at 6 Weeks vs 2.5 mg Injection at Baseline and 6 Weeks; Comparison of the reduction in central subfield thickening in the 1.25mg injection at baseline and at 6 weeks treatment group with the 2.5mg injection at baseline and 6 weeks treatment group at the 6 week visit; Test type: Superiority or Other; p = 0.49, Least squares regression — Adjusted for baseline values
Statistical Analysis 5: Comparison: 1.25 mg Injection at Baseline and at 6 Weeks vs 2.5 mg Injection at Baseline and 6 Weeks; Comparison of the reduction in central subfield thickening in the 1.25mg injection at baseline and at 6 weeks treatment group with the 2.5mg injection at baseline and 6 weeks treatment group at the 9 week visit; Test type: Superiority or Other; p = 0.45, Least squares regression — Adjusted for baseline values
Statistical Analysis 6: Comparison: 1.25 mg Injection at Baseline and at 6 Weeks vs 2.5 mg Injection at Baseline and 6 Weeks; Comparison of the reduction in central subfield thickening in the 1.25mg injection at baseline and at 6 weeks treatment group with the 2.5mg injection at baseline and 6 weeks treatment group at the 12 week visit; Test type: Superiority or Other; p = 0.90, Least squares regression; Adjusted for baseline values

2. Secondary Outcome: Change in Visual Acuity Letter Score From Baseline Over All All Study Visits
Description: Change in visual acuity letter score as measured using an electronic visual acuity testing machine based on the electronic Early Treatment for Diabetic Retinopathy Study(E-ETDRS) technique. At baseline and at each follow up visit, best corrected visual acuity was measured at 3 meters by a certified tester using an electronic procedure based on the E-ETDRS method. Letter score best value = 97 and worst value = 0; positive change represents an improvement in letter score.
Time Frame: Baseline to 3,6,9, and 12 weeks
Measure: Median (Inter-Quartile Range); unit: letters
Arm/Group | Laser at Baseline | 1.25 mg Injection at Baseline and at 6 Weeks | 2.5 mg Injection at Baseline and 6 Weeks | 1.25 mg Injection at Baseline Only | 1.25 mg Injection at Baseline, Laser at 3w + 1.25 mg Inj at 3w
Number analyzed (Participants) | 19 | 22 | 24 | 22 | 22
letters
  3 Weeks | -2 [-7 to 3] | 5 [-1 to 8] | 6 [1 to 9] | 2 [0 to 7] | 0 [-6 to 6]
  6 Weeks | 1 [-6 to 6] | 5 [-2 to 12] | 6 [2 to 11] | 3 [-2 to 6] | 0 [-4 to 6]
  9 Weeks | 3 [-5 to 6] | 7 [2 to 10] | 8 [3 to 12] | 1 [-3 to 5] | -2 [-5 to 11]
  12 Weeks | -1 [-6 to 5] | 5 [1 to 12] | 7 [4 to 11] | 4 [-3 to 7] | 0 [-5 to 8]
Statistical Analysis 1: Comparison: 1.25 mg Injection at Baseline and at 6 Weeks vs 2.5 mg Injection at Baseline and 6 Weeks; Comparison of improvement in visual acuity between the 1.25mg injection at baseline and at 6 weeks treatment group and the 2.5mg injection at baseline and 6 weeks treatment group at the 3 week visit; Test type: Superiority or Other; p = 0.42, Least squares regression; Adjusted for baseline values
Statistical Analysis 2: Comparison: 1.25 mg Injection at Baseline and at 6 Weeks vs 2.5 mg Injection at Baseline and 6 Weeks; Comparison of improvement in visual acuity between the 1.25mg injection at baseline and at 6 weeks treatment group and the 2.5mg injection at baseline and 6 weeks treatment group at the 6 week visit; Test type: Superiority or Other; p = 0.67, Least squares regression; Adjusted for baseline values
Statistical Analysis 3: Comparison: 1.25 mg Injection at Baseline and at 6 Weeks vs 2.5 mg Injection at Baseline and 6 Weeks; Comparison of improvement in visual acuity between the 1.25mg injection at baseline and at 6 weeks treatment group and the 2.5mg injection at baseline and 6 weeks treatment group at the 9 week visit; Test type: Superiority or Other; p = 0.48, Least squares regression; Adjusted for baseline values
Statistical Analysis 4: Comparison: 1.25 mg Injection at Baseline and at 6 Weeks vs 2.5 mg Injection at Baseline and 6 Weeks; Comparison of improvement in visual acuity between the 1.25mg injection at baseline and at 6 weeks treatment group and the 2.5mg injection at baseline and 6 weeks treatment group at the 12 week visit; Test type: Superiority or Other; p = 0.82, Least squares regression
Statistical Analysis 5: Comparison: Laser at Baseline vs 1.25 mg Injection at Baseline and at 6 Weeks; Comparison of improvement in visual acuity through the 12 week visit between the laser only treatment group and the 1.25mg injection at baseline and at 6 weeks treatment group; Test type: Superiority or Other; p = 0.01, Least squares regression; Adjusted for baseline values
Statistical Analysis 6: Comparison: Laser at Baseline vs 2.5 mg Injection at Baseline and 6 Weeks; Comparison of improvement in visual acuity through the 12 week visit between the laser only treatment group and the 2.5mg injection at baseline and at 6 weeks treatment group; Test type: Superiority or Other; p = 0.003, Least squares regression; Adjusted for baseline values

3. Primary Outcome: Percentage of Participants With <250 Microns or ≥ 50% Reduction in Retinal Thickening From Baseline Over All Study Visits
Description: Central subfield retinal thickness measured on Optical Coherence Tomography (OCT). OCT images were obtained at each visit following pupil dilation by a certified operator using the OCT3 machine (Carl Zeiss Meditec Inc., Dublin, CA). Scans were 6 mm length and included the 6 radial line pattern for quantitative measures and the cross hair pattern (6-12 to 9-3 o'clock) for qualitative assessment of retinal morphology. The OCT scans were sent to the DRCR.net Reading Center for grading.
Time Frame: Baseline to 3,6,9, and 12 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Laser at Baseline | 1.25 mg Injection at Baseline and at 6 Weeks | 2.5 mg Injection at Baseline and 6 Weeks | 1.25 mg Injection at Baseline Only | 1.25 mg Injection at Baseline, Laser at 3w + 1.25 mg Inj at 3w
Number analyzed (Participants) | 19 | 22 | 24 | 22 | 22
percentage of participants
  3 Weeks | 11 | 37 | 38 | 10 | 25
  6 Weeks | 17 | 30 | 22 | 19 | 25
  9 Weeks | 19 | 38 | 22 | 10 | 37
  12 Weeks | 21 | 33 | 33 | 14 | 25

4. Secondary Outcome: Distribution of Change in Visual Acuity Over All Study Visits
Description: Visual acuity letter score as measured using an electronic visual acuity testing machine based on the electronic Early Treatment for Diabetic Retinopathy Study(E-ETDRS) technique. At baseline and at each follow up visit, best corrected visual acuity was measured at 3 meters by a certified tester using an electronic procedure based on the E-ETDRS method. Letter score best value = 97 and worst value = 0; an increase in a letter score by 10 is considered clinically significant.
Time Frame: Baseline to 3,6,9, and 12 weeks
Measure: Number; unit: participants
Arm/Group | Laser at Baseline | 1.25 mg Injection at Baseline and at 6 Weeks | 2.5 mg Injection at Baseline and 6 Weeks | 1.25 mg Injection at Baseline Only | 1.25 mg Injection at Baseline, Laser at 3w + 1.25 mg Inj at 3w
Number analyzed (Participants) | 19 | 22 | 24 | 22 | 22
participants
  ≥ 10 letter improvement at 3 Weeks | 1 | 4 | 4 | 2 | 2
  ≥ 10 letters worse at 3 Weeks | 1 | 1 | 0 | 1 | 0
  ≥ 10 letter improvement at 6 Weeks | 2 | 7 | 7 | 3 | 3
  ≥ 10 letters worse at 6 Weeks | 2 | 0 | 1 | 1 | 4
  ≥ 10 letter improvement at 9 Weeks | 3 | 6 | 9 | 3 | 5
  ≥ 10 letters worse at 9 Weeks | 1 | 1 | 0 | 0 | 2
  ≥ 10 letter improvement at 12 Weeks | 3 | 7 | 6 | 2 | 4
  ≥ 10 letters worse at 12 Weeks | 1 | 1 | 0 | 2 | 2

5. Other Pre Specified Outcome: Change in Central Subfield Thickness in Bevacizumab Groups From Baseline to 3 Weeks According to Baseline Central Subfield Thickness
Description: Pooled Bevacizumab groups include the following treatment groups: 1.25mg at baseline and at 6 weeks, 2.5mg at baseline and at 6 weeks, 1.25mg at baseline only, and 1.25mg at baseline and 6 weeks plus laser at 3 weeks. Negative values represent a reduction in central subfield thickness. The 4 bevacizumab groups (N=87) were pooled to compare differences in response at 3 weeks among subgroups of interest. The pooled Bevacizumab treatment group will be the only group/arm that has values, all other treatment groups/arms will have a null value for this outcome measure.
Time Frame: Baseline to 3 Weeks
Measure: Median (Inter-Quartile Range); unit: microns
Groups:
- Pooled Bevacizumab Groups: Pooled Bevacizumab group includes the following treatment groups: 1.25mg at baseline and at 6 weeks; 2.5mg at baseline and at 6 weeks; 1.25mg at baseline only; and 1.25mg at baseline and 6 weeks plus laser at 3 weeks.
Arm/Group | Pooled Bevacizumab Groups
Number analyzed (Participants) | 87
microns
  <400 microns | -3 [-49 to 13]
  ≥400 microns | -102 [-145 to -6]
Statistical Analysis 1: Comparison: Pooled Bevacizumab Groups; Comparison of central subfield thickness (microns) change from baseline to the 3 week visit between eyes that had baseline central subfield thickness of <400 microns compared to those that had baseline central subfield thickness of ≥400 microns. Eyes included all of those from the pooled Bevacizumab group; Test type: Superiority or Other; p < 0.0001, Least squares regression; Adjusted for baseline values

6. Other Pre Specified Outcome: Change in Central Subfield Thickness in Bevacizumab Groups From Baseline to 3 Weeks According to Baseline Visual Acuity Letter Score
Description: Pooled Bevacizumab group includes the following treatment groups: 1.25mg at baseline and at 6 weeks, 2.5mg at baseline and at 6 weeks, 1.25mg at baseline only, and 1.25mg at baseline and 6 weeks plus laser at 3 weeks. Negative values represent a reduction in central subfield thickness. The 4 bevacizumab groups (N=87) were pooled to compare differences in response at 3 weeks among subgroups of interest. The pooled Bevacizumab treatment group will be the only group/arm that has values, all other treatment groups/arms will have a null value for this outcome measure.
Time Frame: Baseline to 3 Weeks
Measure: Median (Inter-Quartile Range); unit: microns
Arm/Group | Pooled Bevacizumab Groups
Number analyzed (Participants) | 87
microns
  <65 letters | -35 [-130 to 5]
  ≥65 letters | -28 [-102 to 13]
Statistical Analysis 1: Comparison: Pooled Bevacizumab Groups; Comparison of central subfield thickness (microns) change from baseline to the 3 week visit between eyes that had baseline visual acuity letter score that was <65 letters compared to those that had baseline visual acuity letter score that was ≥65 letters. Eyes included all of those from the pooled Bevacizumab group; Test type: Superiority or Other; p = 0.31, Least squares regression; Adjusted for baseline score

7. Other Pre Specified Outcome: Change in Central Subfield Thickness in Bevacizumab Groups From Baseline to 3 Weeks According to Age at Baseline
Description: as for outcome 6
Time Frame: Baseline to 3 Weeks
Measure: Median (Inter-Quartile Range); unit: microns
Arm/Group | Pooled Bevacizumab Groups
Number analyzed (Participants) | 87
microns
  ≤66 years | -45 [-131 to 5]
  >66 years | -16 [-107 to 6]
Statistical Analysis 1: Comparison: Pooled Bevacizumab Groups; Comparison of central subfield thickness (microns) change from baseline to the 3 week visit between those that were ≤66 years old compared to those that were >66 years old at baseline. Eyes included all of those from the pooled Bevacizumab group; Test type: Superiority or Other; p = 0.44, Least squares regression

8. Other Pre Specified Outcome: Change in Central Subfield Thickness in Bevacizumab Groups From Baseline to 3 Weeks According to Gender
Description: as for outcome 6
Time Frame: Baseline to 3 Weeks
Measure: Median (Inter-Quartile Range); unit: microns
Arm/Group | Pooled Bevacizumab Groups
Number analyzed (Participants) | 87
microns
  Female | -28 [-115 to 6]
  Male | -35 [-105 to 5]
Statistical Analysis 1: Comparison: Pooled Bevacizumab Groups; Comparison of central subfield thickness (microns) change from baseline to the 3 week visit between females and males. Eyes included all of those from the pooled Bevacizumab group; Test type: Superiority or Other; p = 0.55, Least squares regression

9. Other Pre Specified Outcome: Change in Central Subfield Thickness in Bevacizumab Groups From Baseline to 3 Weeks According to History of Treatment for Diabetic Macular Edema at Baseline
Description: as for outcome 6
Time Frame: Baseline to 3 Weeks
Measure: Median (Inter-Quartile Range); unit: microns
Arm/Group | Pooled Bevacizumab Groups
Number analyzed (Participants) | 87
microns
  No | -40 [-141 to -3]
  Yes | -29 [-102 to 7]
Statistical Analysis 1: Comparison: Pooled Bevacizumab Groups; Comparison of central subfield thickness (microns) change from baseline to the 3 week visit between eyes that had no history of treatment for diabetic macular edema compared to those that had history or treatment for diabetic macular edema. Eyes included all of those from the pooled Bevacizumab group; Test type: Superiority or Other; p = 0.16, Least squares regression; Adjusted for baseline values

10. Other Pre Specified Outcome: Change in Central Subfield Thickness in Bevacizumab Groups From Baseline to 3 Weeks According to Retinopathy Severity at Baseline
Description: Pooled Bevacizumab group includes treatment groups: 1.25mg at baseline and at 6 weeks, 2.5mg at baseline and at 6 weeks, 1.25mg at baseline only, and 1.25mg at baseline and 6 weeks + laser at 3 weeks. Negative values represent a reduction in central subfield thickness. The 4 bevacizumab groups (N=87) were pooled to compare differences in response at 3 weeks among subgroups of interest. Retinopathy severity based on investigator discretion on clinical examination.
Time Frame: baseline to 3 Weeks
Measure: Median (Inter-Quartile Range); unit: microns
Arm/Group | Pooled Bevacizumab Groups
Number analyzed (Participants) | 87
microns
  <Severe nonproliferative diabetic retinopathy | -31 [-115 to 6]
  Proliferative diabetic retinopathy or severe NPDR | -31 [-105 to 13]
Statistical Analysis 1: Comparison: Pooled Bevacizumab Groups; Comparison of central subfield thickness (microns) change from baseline to the 3 week visit between eyes that had baseline retinopathy severity that was <severe nonproliferative diabetic retinopathy (NPDR) compared to those that had baseline retinopathy severity that was proliferative diabetic retinopathy or severe NPDR. Eyes included all of those from the pooled Bevacizumab group; Test type: Superiority or Other; p = 0.53, Least squares regression

11. Other Pre Specified Outcome: Change in Central Subfield Thickness in Bevacizumab Groups From Baseline to 3 Weeks According to Clinical Diabetic Macular Edema Characterization at Baseline
Description: as for outcome 6
Time Frame: baseline to 3 Weeks
Measure: Median (Inter-Quartile Range); unit: microns
Arm/Group | Pooled Bevacizumab Groups
Number analyzed (Participants) | 87
microns
  Typical/Predominantly Focal | -13 [-67 to -2]
  Neither Predominantly Focal or Diffuse | -8 [-32 to 20]
  Typical/Predominantly Diffuse | -82 [-139 to 5]
Statistical Analysis 1: Comparison: Pooled Bevacizumab Groups; Comparison of central subfield thickness (microns) change from baseline to the 3 week visit between eyes that had baseline clinical diabetic macular edema characterized as typical/predominantly focal, neither predominantly focal or diffuse, or typical/predominantly diffuse. Eyes included all of those from the pooled Bevacizumab group; Test type: Superiority or Other; p = 0.93, Least squares regression; Adjusted for baseline values

12. Other Pre Specified Outcome: Change in Central Subfield Thickness in Bevacizumab Groups From Baseline to 3 Weeks According to Subretinal Fluid Presence at Baseline
Description: as for outcome 6
Time Frame: baseline to 3 Weeks
Measure: Median (Inter-Quartile Range); unit: microns
Arm/Group | Pooled Bevacizumab Groups
Number analyzed (Participants) | 87
microns
  Definite/Questionable | -35 [-131 to 24]
  No Evidence | -29 [-102 to 3]
Statistical Analysis 1: Comparison: Pooled Bevacizumab Groups; Comparison of central subfield thickness (microns) change from baseline to the 3 week visit between eyes that had baseline subretinal fluid that was definite/questionable compared to eyes that had no evidence of subretinal fluid at baseline. Eyes included all of those from the pooled Bevacizumab group; Test type: Superiority or Other; p = 0.52, Least squares regression; Adjusted for baseline values

13. Other Pre Specified Outcome: Change in Visual Acuity (Letters) in Bevacizumab Groups From Baseline to 3 Weeks According to Central Subfield Thickness at Baseline
Description: Pooled Bevacizumab group includes the following treatment groups: 1.25mg at baseline and at 6 weeks, 2.5mg at baseline and at 6 weeks, 1.25mg at baseline only, and 1.25mg at baseline and 6 weeks plus laser at 3 weeks. The 4 bevacizumab groups (N=87) were pooled to compare differences in response at 3 weeks among subgroups of interest. The pooled Bevacizumab treatment group will be the only group/arm that has values, all other treatment groups/arms will have a null value for this outcome measure. Positive values represent an improvement in letter score.
Time Frame: baseline to 3 Weeks
Measure: Median (Inter-Quartile Range); unit: letters
Arm/Group | Pooled Bevacizumab Groups
Number analyzed (Participants) | 87
letters
  <400 microns | 1 [-2 to 8]
  ≥400 microns | 5 [0 to 8]
Statistical Analysis 1: Comparison: Pooled Bevacizumab Groups; Comparison of change in visual acuity letter score from baseline to the 3 week visit between eyes that had baseline central subfield thickness of <400 microns compared to eyes that had baseline central subfield thickness of ≥400 microns. Eyes included all of those from the pooled Bevacizumab group; Test type: Superiority or Other; p = 0.22, Least squares regression; Adjusted for baseline values

14. Other Pre Specified Outcome: Change in Visual Acuity (Letters) in Bevacizumab Groups From Baseline to 3 Weeks According to Visual Acuity at Baseline
Description: as for outcome 13
Time Frame: baseline to 3 Weeks
Measure: Median (Inter-Quartile Range); unit: letters
Arm/Group | Pooled Bevacizumab Groups
Number analyzed (Participants) | 87
letters
  <65 letters | 3 [0 to 9]
  ≥65 letters | 1 [-3 to 7]
Statistical Analysis 1: Comparison: Pooled Bevacizumab Groups; Comparison of change in visual acuity letter score from baseline to the 3 week visit between eyes that had a baseline visual acuity letter score of <65 letters compared to eyes that had baseline visual acuity letter score of ≥65 letters. Eyes included all of those from the pooled Bevacizumab group; Test type: Superiority or Other; p = 0.006, Least squares regression; Adjusted for baseline values

15. Other Pre Specified Outcome: Change in Visual Acuity (Letters) in Bevacizumab Groups From Baseline to 3 Weeks According to Age at Baseline
Description: as for outcome 13
Time Frame: baseline to 3 Weeks
Measure: Median (Inter-Quartile Range); unit: letters
Arm/Group | Pooled Bevacizumab Groups
Number analyzed (Participants) | 87
letters
  ≤66 years | 4 [-1 to 8]
  >66 years | 2 [0 to 8]
Statistical Analysis 1: Comparison: Pooled Bevacizumab Groups; Comparison of change in visual acuity letter score from baseline to the 3 week visit between eyes that were ≤66 years old at baseline compared to eyes that were >66 years old at baseline. Eyes included all of those from the pooled Bevacizumab group; Test type: Superiority or Other; p = 0.23, Least squares regression

16. Other Pre Specified Outcome: Change in Visual Acuity (Letters) in Bevacizumab Groups From Baseline to 3 Weeks According to Gender
Description: as for outcome 13
Time Frame: baseline to 3 Weeks
Measure: Median (Inter-Quartile Range); unit: letters
Arm/Group | Pooled Bevacizumab Groups
Number analyzed (Participants) | 87
letters
  Female | 3 [0 to 8]
  Male | 3 [-1 to 7]
Statistical Analysis 1: Comparison: Pooled Bevacizumab Groups; Comparison of change in visual acuity letter score from baseline to the 3 week visit between females and males. Eyes included all of those from the pooled Bevacizumab group; Test type: Superiority or Other; p = 0.37, Least squares regression

17. Other Pre Specified Outcome: Change in Visual Acuity (Letters) in Bevacizumab Groups From Baseline to 3 Weeks According to History of Treatment for Diabetic Macular Edema
Description: as for outcome 13
Time Frame: baseline to 3 Weeks
Measure: Median (Inter-Quartile Range); unit: letters
Arm/Group | Pooled Bevacizumab Groups
Number analyzed (Participants) | 87
letters
  No | 5 [-1 to 8]
  Yes | 2 [-1 to 8]
Statistical Analysis 1: Comparison: Pooled Bevacizumab Groups; Comparison of change in visual acuity letter score from baseline to the 3 week visit between eyes that did not have a prior history of treatment for diabetic macular edema compared to eyes that did have a prior history of treatment for diabetic macular edema. Eyes included all of those from the pooled Bevacizumab group; Test type: Superiority or Other; p = 0.04, Least squares regression

18. Other Pre Specified Outcome: Change in Visual Acuity (Letters) in Bevacizumab Groups From Baseline to 3 Weeks According to Retinopathy Severity at Baseline
Description: as for outcome 13
Time Frame: baseline to 3 Weeks
Measure: Median (Inter-Quartile Range); unit: letters
Arm/Group | Pooled Bevacizumab Groups
Number analyzed (Participants) | 87
letters
  <Severe nonproliferative diabetic retinopathy | 3 [0 to 8]
  Proliferative diabetic retinopathy or severe NPDR | 1 [-3 to 7]
Statistical Analysis 1: Comparison: Pooled Bevacizumab Groups; Comparison of change in visual acuity letter score from baseline to the 3 week visit between eyes that had a baseline retinopathy severity of <severe nonproliferative diabetic retinopathy (NPDR) compared to eyes that had baseline retinopathy severity of proliferative diabetic retinopathy or severe NPDR. Eyes included all of those from the pooled Bevacizumab group; Test type: Superiority or Other; p = 0.38, Least squares regression

19. Other Pre Specified Outcome: Change in Visual Acuity (Letters) in Bevacizumab Groups From Baseline to 3 Weeks According to Clinical Diabetic Macular Edema Characterization at Baseline
Description: as for outcome 13
Time Frame: baseline to 3 Weeks
Measure: Median (Inter-Quartile Range); unit: letters
Arm/Group | Pooled Bevacizumab Groups
Number analyzed (Participants) | 87
letters
  Typical/Predominantly Focal | 7 [0 to 9]
  Neither Predominantly Focal or Diffuse | 0 [-5 to 5]
  Typical/Predominantly Diffuse | 3 [0 to 8]
Statistical Analysis 1: Comparison: Pooled Bevacizumab Groups; Comparison of change in visual acuity letter score from baseline to the 3 week visit between eyes that had a baseline clinical diabetic macular edema (DME) characterization of typical/predominantly focal compared to neither predominantly focal or diffuse characterization at baseline and compared to typical/predominantly diffuse characterization at baseline. Eyes included all of those from the pooled Bevacizumab group; Test type: Superiority or Other; p = 0.45, Least squares regression

20. Other Pre Specified Outcome: Change in Visual Acuity (Letters) in Bevacizumab Groups From Baseline to 3 Weeks According to Subretinal Fluid Presence at Baseline
Description: as for outcome 13
Time Frame: baseline to 3 Weeks
Measure: Median (Inter-Quartile Range); unit: letters
Arm/Group | Pooled Bevacizumab Groups
Number analyzed (Participants) | 87
letters
  Definite/Questionable | 6 [3 to 11]
  No Evidence | 1 [-1 to 7]
Statistical Analysis 1: Comparison: Pooled Bevacizumab Groups; Comparison of change in visual acuity letter score from baseline to the 3 week visit between eyes that had a baseline subretinal fluid presence that was definite/questionable compared to eyes that there was no evidence of subretinal fluid at baseline. Eyes included all of those from the pooled Bevacizumab group; Test type: Superiority or Other; p = 0.06, Least squares regression

21. Other Pre Specified Outcome: Change in Central Subfield Thickness From 3 to 6 Weeks Among Eyes That Received 1.25mg Injection Only and Had a >11% Decrease in Change of Central Subfield Thickness From Baseline to 3 Weeks
Description: The 1.25mg Bevacizumab groups include the following treatment groups: 1.25mg at baseline and 6 weeks; and 1.25mg at baseline only. Duration of effect of Bevacizumab was based on additional improvement versus maintained improvement versus worsening within 3 to 6 weeks. Change in central subfield thickness was categorized according to whether it exceeded 11%, the reliability limit for real change determined in the DRCR.net paper, Reproducibility of macular thickness and volume using Zeiss optical coherence tomography in patients with diabetic macular edema.Ophthalmology 2007;114:1520-25.
Time Frame: 3 to 6 Weeks
Measure: Number; unit: Participants
Groups:
- Pooled 1.25mg Initial Bevacizumab Injection Groups: The following are the treatment groups included in the Pooled 1.25mg Bevacizumab Groups: 1.25mg at baseline and 6 weeks; and 1.25mg at baseline only
Arm/Group | Pooled 1.25mg Initial Bevacizumab Injection Groups
Number analyzed (Participants) | 14
Participants
  >11% Decreased Change from 3 Weeks to 6 Weeks | 1
  Within ± 11% Change from 3 Weeks to 6 Weeks | 11
  >11% Increased Change from 3 Weeks to 6 Weeks | 2

22. Other Pre Specified Outcome: Change in Central Subfield Thickness From 3 to 6 Weeks Among Eyes That Received 1.25mg Injection Only and Had Within a ±11% Change of Central Subfield Thickness From Baseline to 3 Weeks
Description: The 1.25mg bevacizumab groups include the following treatment groups: 1.25mg at baseline and 6 weeks; and 1.25mg at baseline only. Change in central subfield thickness was categorized according to whether it exceeded 11%, the reliability limit for real change determined in another Diabetic Retinopathy Clinical Research Network study 16. The pooled 1.25mg bevacizumab treatment group will be the only group/arm that has values, all other treatment groups/arms will have a null value for this outcome measure.
Time Frame: 3 to 6 Weeks
Measure: Number; unit: participants
Arm/Group | Pooled 1.25mg Initial Bevacizumab Injection Groups
Number analyzed (Participants) | 22
participants
  >11% Decreased Change from 3 Weeks to 6 Weeks | 2
  Within ± 11% Change from 3 Weeks to 6 Weeks | 16
  >11% Increased Change from 3 Weeks to 6 Weeks | 4

23. Other Pre Specified Outcome: Change in Central Subfield Thickness From 3 to 6 Weeks Among Eyes That Received 1.25mg Injection Only and Had a >11% Increase in Change of Central Subfield Thickness From Baseline to 3 Weeks
Description: as for outcome 22
Time Frame: 3 to 6 Weeks
Measure: Number; unit: Participants
Arm/Group | Pooled 1.25mg Initial Bevacizumab Injection Groups
Number analyzed (Participants) | 2
Participants
  >11% Decreased Change from 3 Weeks to 6 Weeks | 1
  Within ± 11% Change from 3 Weeks to 6 Weeks | 1
  >11% Increased Change from 3 Weeks to 6 Weeks | 0

24. Other Pre Specified Outcome: Change in Central Subfield Thickness From 3 to 6 Weeks Among Eyes That Received 2.5mg Bevacizumab and Had a >11% Decrease in Change of Central Subfield Thickness From Baseline to 3 Weeks
Description: The 2.5mg bevacizumab treatment group received an injection at both baseline and at 6 weeks. Change in central subfield thickness was categorized according to whether it exceeded 11%, the reliability limit for real change determined in another Diabetic Retinopathy Clinical Research Network study 16. The 2.5mg bevacizumab treatment group will be the only group/arm that has values, all other treatment groups/arms will have a null value for this outcome measure.
Time Frame: 3 to 6 Weeks
Measure: Number; unit: Participants
Arm/Group | 2.5 mg Injection at Baseline and 6 Weeks
Number analyzed (Participants) | 13
Participants
  >11% Decreased Change from 3 Weeks to 6 Weeks | 0
  Within ± 11% Change from 3 Weeks to 6 Weeks | 9
  >11% Increased Change from 3 Weeks to 6 Weeks | 4

25. Other Pre Specified Outcome: Change in Central Subfield Thickness From 3 to 6 Weeks Among Eyes That Received 2.5mg Bevacizumab and Had Within a ±11% Change in Central Subfield Thickness From Baseline to 3 Weeks
Description: as for outcome 24
Time Frame: 3 to 6 Weeks
Measure: Number; unit: participants
Arm/Group | 2.5 mg Injection at Baseline and 6 Weeks
Number analyzed (Participants) | 10
participants
  >11% Decreased Change from 3 Weeks to 6 Weeks | 0
  Within ± 11% Change from 3 Weeks to 6 Weeks | 9
  >11% Increased Change from 3 Weeks to 6 Weeks | 1

26. Other Pre Specified Outcome: Change in Central Subfield Thickness From 3 to 6 Weeks Among Eyes That Received 2.5mg Bevacizumab and Had a >11% Increase in Change of Central Subfield Thickness From Baseline to 3 Weeks
Description: as for outcome 24
Time Frame: 3 to 6 Weeks
Population: There were no participants with a change in central subfield thickness from 3 to 6 weeks in this treatment group that had a >11% increase in change of central subfield thickness from baseline to 3 weeks.
Arm/Group | 2.5 mg Injection at Baseline and 6 Weeks
Number analyzed (Participants) | 0

27. Other Pre Specified Outcome: Change in Central Subfield Thickness From 3 to 6 Weeks Among Eyes That Received 1.25mg Bevacizumab at 6 Weeks and Had a >11% Decrease in Change of Central Subfield Thickness From 6 Weeks to 9 Weeks
Description: The 1.25mg bevacizumab treatment group received an injection at both baseline and at 6 weeks. Change in central subfield thickness was categorized according to whether it exceeded 11%, the reliability limit for real change determined in another Diabetic Retinopathy Clinical Research Network study 16. The 1.25mg bevacizumab treatment group will be the only group/arm that has values, all other treatment groups/arms will have a null value for this outcome measure.
Time Frame: 3 to 9 weeks
Measure: Number; unit: participants
Arm/Group | 1.25 mg Injection at Baseline and at 6 Weeks
Number analyzed (Participants) | 7
participants
  >11% Decreased Change from 9 Weeks to 12 Weeks | 0
  Within ± 11% Change from 9 Weeks to 12 Weeks | 4
  >11% Increased Change from 9 Weeks to 12 Weeks | 3

28. Other Pre Specified Outcome: Change in Central Subfield Thickness From 3 to 6 Weeks Among Eyes That Received 1.25mg Bevacizumab at 6 Weeks and Had Within ±11% Change of Central Subfield Thickness From 6 Weeks to 9 Weeks
Description: as for outcome 27
Time Frame: 3 to 9 weeks
Measure: Number; unit: participants
Arm/Group | 1.25 mg Injection at Baseline and at 6 Weeks
Number analyzed (Participants) | 9
participants
  >11% Decreased Change from 9 Weeks to 12 Weeks | 1
  Within ± 11% Change from 9 Weeks to 12 Weeks | 6
  >11% Increased Change from 9 Weeks to 12 Weeks | 2

29. Other Pre Specified Outcome: Change in Central Subfield Thickness From 3 to 6 Weeks Among Eyes That Received 1.25mg Bevacizumab at 6 Weeks and Had a >11% Increase in Change of Central Subfield Thickness From 6 Weeks to 9 Weeks
Description: as for outcome 27
Time Frame: 3 to 9 weeks
Measure: Number; unit: participants
Arm/Group | 1.25 mg Injection at Baseline and at 6 Weeks
Number analyzed (Participants) | 2
participants
  >11% Decreased Change from 9 Weeks to 12 Weeks | 0
  Within ± 11% Change from 9 Weeks to 12 Weeks | 2
  >11% Increased Change from 9 Weeks to 12 Weeks | 0

30. Other Pre Specified Outcome: Change in Central Subfield Thickness From 3 to 6 Weeks Among Eyes That Received 2.5mg Bevacizumab at 6 Weeks and Had a >11% Decrease in Change of Central Subfield Thickness From 6 Weeks to 9 Weeks
Description: as for outcome 24
Time Frame: 3 to 9 weeks
Measure: Number; unit: participants
Arm/Group | 2.5 mg Injection at Baseline and 6 Weeks
Number analyzed (Participants) | 3
participants
  >11% Decreased Change from 9 Weeks to 12 Weeks | 0
  Within ± 11% Change from 9 Weeks to 12 Weeks | 2
  >11% Increased Change from 9 Weeks to 12 Weeks | 1

31. Other Pre Specified Outcome: Change in Central Subfield Thickness From 3 to 6 Weeks Among Eyes That Received 2.5mg Bevacizumab at 6 Weeks and Had Within ±11% Change of Central Subfield Thickness From 6 Weeks to 9 Weeks
Description: as for outcome 24
Time Frame: 3 to 9 weeks
Measure: Number; unit: participants
Arm/Group | 2.5 mg Injection at Baseline and 6 Weeks
Number analyzed (Participants) | 17
participants
  >11% Decreased Change from 9 Weeks to 12 Weeks | 2
  Within ± 11% Change from 9 Weeks to 12 Weeks | 14
  >11% Increased Change from 9 Weeks to 12 Weeks | 1

32. Other Pre Specified Outcome: Change in Central Subfield Thickness From 3 to 6 Weeks Among Eyes That Received 2.5mg Bevacizumab at 6 Weeks and Had Within >11% Increase in Change of Central Subfield Thickness From 6 Weeks to 9 Weeks
Description: as for outcome 24
Time Frame: 3 to 9 weeks
Measure: Number; unit: participants
Arm/Group | 2.5 mg Injection at Baseline and 6 Weeks
Number analyzed (Participants) | 2
participants
  >11% Decreased Change from 9 Weeks to 12 Weeks | 1
  Within ± 11% Change from 9 Weeks to 12 Weeks | 1
  >11% Increased Change from 9 Weeks to 12 Weeks | 0

ADVERSE EVENTS:
Arm/Group | Laser at Baseline | 1.25 mg Injection at Baseline and at 6 Weeks | 2.5 mg Injection at Baseline and 6 Weeks | 1.25 mg Injection at Baseline Only | 1.25 mg Injection at Baseline, Laser at 3w + 1.25 mg Inj at 3w
Serious Adverse Events (participants affected / at risk) | 8/19 | 8/22 | 6/24 | 1/22 | 6/22
Other Adverse Events (participants affected / at risk) | 14/19 | 16/22 | 19/24 | 20/22 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Laser at Baseline (N=19) | 1.25 mg Injection at Baseline and at 6 Weeks (N=22) | 2.5 mg Injection at Baseline and 6 Weeks (N=24) | 1.25 mg Injection at Baseline Only (N=22) | 1.25 mg Injection at Baseline, Laser at 3w + 1.25 mg Inj at 3w (N=22)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Bacterial skin infection (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Cellulitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Cerebrovascular accident (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Congestive cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Death (General disorders) | 1 | 1 | 0 | 0 | 0
Delerium (General disorders) | 0 | 0 | 1 | 0 | 0
Endophthalmitis (General disorders) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Glaucoma (General disorders) | 0 | 0 | 0 | 0 | 1
Hip fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Inadequate control of diabetes mellitus (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Intraventricular haemorrhage (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Metastatic lung cancer (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 3
Pancreatic carcinoma (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Skin ulcer or skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Syncope (General disorders) | 0 | 1 | 0 | 0 | 0
Vitrectomy (General disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Laser at Baseline (N=19) | 1.25 mg Injection at Baseline and at 6 Weeks (N=22) | 2.5 mg Injection at Baseline and 6 Weeks (N=24) | 1.25 mg Injection at Baseline Only (N=22) | 1.25 mg Injection at Baseline, Laser at 3w + 1.25 mg Inj at 3w (N=22)
Abdominal pain (General disorders) | 0 | 1 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 1
Angle Closure Glaucoma (Eye disorders) | 0 | 1 | 0 | 0 | 0
Anorexia (General disorders) | 0 | 0 | 0 | 0 | 1
Anterior chamber cell (Eye disorders) | 0 | 0 | 0 | 0 | 1
Anterior chamber flare (Eye disorders) | 0 | 0 | 0 | 0 | 1
Back injury (General disorders) | 0 | 0 | 1 | 0 | 0
Blepharitis (Eye disorders) | 1 | 2 | 0 | 1 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 1
Cataract nuclear (Eye disorders) | 0 | 2 | 1 | 0 | 0
Cerebrovascular accident (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Conjunctival hemorrhage (Eye disorders) | 0 | 5 | 1 | 6 | 3
Diabetes mellitus (Endocrine disorders) | 0 | 1 | 0 | 0 | 1
Diabetic Retinopathy (Eye disorders) | 0 | 1 | 0 | 0 | 1
Diabetic retinal edema (Eye disorders) | 0 | 5 | 3 | 2 | 1
Diplopia (Eye disorders) | 0 | 2 | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 1 | 0 | 2 | 1
Eye pain (Eye disorders) | 2 | 4 | 5 | 3 | 5
Foreign body sensation in eyes (Eye disorders) | 1 | 0 | 2 | 0 | 2
Gastroenteritis viral (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Headache (General disorders) | 1 | 2 | 0 | 1 | 1
Hypercholesterolemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 2 | 0
Hypertension (Vascular disorders) | 2 | 2 | 2 | 1 | 1
Increased intraocular pressure (Eye disorders) | 0 | 1 | 3 | 3 | 2
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1
Lacrimation increased (Eye disorders) | 1 | 3 | 2 | 2 | 1
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 1 | 0 | 2
Osteomyelitis (General disorders) | 1 | 0 | 0 | 0 | 0
Peripheral vascular disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Tooth abcess (General disorders) | 0 | 2 | 0 | 0 | 0
Vision blurred (Eye disorders) | 5 | 6 | 5 | 5 | 5
Visual acuity reduced (Eye disorders) | 2 | 4 | 0 | 1 | 0
Visual disturbance (Eye disorders) | 0 | 0 | 4 | 2 | 1
Vitreous floaters (Eye disorders) | 0 | 7 | 8 | 1 | 3
Vitreous hemorrhage (Eye disorders) | 0 | 1 | 5 | 3 | 2
anxiety (General disorders) | 0 | 0 | 0 | 1 | 1
arthralgia (General disorders) | 0 | 0 | 1 | 0 | 0
asbestosis (General disorders) | 0 | 0 | 0 | 0 | 1
autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
back pain (General disorders) | 0 | 1 | 0 | 0 | 1
benign breast neoplasm (General disorders) | 0 | 0 | 0 | 1 | 0
blister (General disorders) | 0 | 0 | 0 | 1 | 0
blood creatine increased (General disorders) | 0 | 0 | 0 | 0 | 1
blood glucose decreased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
blood potassium increased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
breast cancer (General disorders) | 0 | 0 | 0 | 1 | 0
cataract (Eye disorders) | 1 | 1 | 0 | 1 | 1
cataract cortical (Eye disorders) | 0 | 1 | 0 | 0 | 0
cataract operation (Eye disorders) | 0 | 0 | 0 | 1 | 1
cataract operation complication (Eye disorders) | 0 | 0 | 0 | 0 | 1
cataract subcapsular (Eye disorders) | 1 | 0 | 0 | 1 | 1
caugh (General disorders) | 0 | 1 | 0 | 0 | 0
chalazion (General disorders) | 0 | 0 | 0 | 0 | 1
chest pain (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
chronic obstructive pulmonary disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
colon cancer (General disorders) | 0 | 0 | 1 | 0 | 0
conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 1 | 0
conjunctivitis viral (Eye disorders) | 0 | 0 | 0 | 0 | 1
constipation (General disorders) | 1 | 0 | 0 | 0 | 0
corneal abrasion (Eye disorders) | 0 | 1 | 0 | 0 | 1
corneal oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1
deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1
desemets membrane disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1
diabetes mellitus inadequate control (Endocrine disorders) | 0 | 1 | 0 | 0 | 1
dizziness (General disorders) | 0 | 0 | 1 | 1 | 1
dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 1
epistaxis (General disorders) | 0 | 0 | 1 | 0 | 0
eye inflammation (Eye disorders) | 0 | 1 | 0 | 0 | 0
eye pruritus (Eye disorders) | 0 | 1 | 1 | 1 | 1
eyelid oedema (Eye disorders) | 0 | 1 | 1 | 0 | 1
eyelid pain (Eye disorders) | 1 | 0 | 1 | 0 | 0
eyelid ptsosis (Eye disorders) | 1 | 0 | 0 | 1 | 0
fall (General disorders) | 0 | 0 | 1 | 0 | 0
foreign body in eye (Eye disorders) | 0 | 0 | 0 | 1 | 0
fungal skin infection (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
gastrooespohageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
haematochezia (General disorders) | 0 | 0 | 0 | 1 | 0
haemoglobin decreased (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
heart rate irregular (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
herpes zoster (General disorders) | 1 | 0 | 0 | 0 | 0
hyperkalaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0
hypoglycaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
injection site irritaion (Eye disorders) | 0 | 0 | 0 | 1 | 0
insomnia (General disorders) | 0 | 0 | 1 | 0 | 0
intervertebral disc protrusion (General disorders) | 1 | 0 | 0 | 0 | 0
joint dislocation (General disorders) | 1 | 0 | 0 | 0 | 0
keratoconjunctivitis sicca (Eye disorders) | 1 | 1 | 0 | 1 | 1
leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
localised infection (General disorders) | 1 | 0 | 0 | 0 | 1
macular oedema (Eye disorders) | 1 | 0 | 1 | 0 | 1
maculopathy (Eye disorders) | 1 | 1 | 2 | 1 | 0
nasopharyngitis (General disorders) | 1 | 0 | 3 | 0 | 0
nausea (General disorders) | 0 | 1 | 1 | 0 | 1
nerve injury (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
oedema peripheral (Eye disorders) | 1 | 1 | 0 | 0 | 0
optic nerve cupping (Eye disorders) | 1 | 0 | 0 | 0 | 0
pain in extremity (General disorders) | 0 | 0 | 0 | 1 | 1
periorbital haematoma (Eye disorders) | 1 | 0 | 0 | 0 | 0
peritonitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
pharyngolaryngeal pain (General disorders) | 0 | 0 | 0 | 0 | 1
photophobia (Eye disorders) | 0 | 1 | 0 | 0 | 0
photopsia (Eye disorders) | 0 | 1 | 1 | 1 | 0
posterior capsule opacification (Eye disorders) | 0 | 0 | 0 | 1 | 1
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
protein urine present (General disorders) | 1 | 0 | 0 | 0 | 0
pruritus (General disorders) | 0 | 1 | 0 | 0 | 0
pterygium (Eye disorders) | 0 | 0 | 0 | 1 | 0
punctate keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
reading disorder (General disorders) | 0 | 0 | 0 | 0 | 1
renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0
renal failure chronic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
respiratory tract congestion (General disorders) | 0 | 0 | 1 | 0 | 0
retinal degeneration (Eye disorders) | 0 | 0 | 1 | 0 | 0
retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1
retinal exudates (Eye disorders) | 0 | 0 | 0 | 0 | 1
retinal laser coagulation (Eye disorders) | 0 | 0 | 1 | 0 | 0
retinal neovascularisation (Eye disorders) | 0 | 0 | 1 | 0 | 0
retinal oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0
retinal telagiectasia (Eye disorders) | 0 | 0 | 0 | 1 | 0
rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
rhinitis allergic (General disorders) | 0 | 1 | 0 | 1 | 0
sinusitis (General disorders) | 0 | 0 | 0 | 0 | 1
skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
skin lesion excision (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
swollen tongue (General disorders) | 0 | 0 | 1 | 0 | 0
trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
upper respiratory tract infection (General disorders) | 0 | 1 | 1 | 0 | 0
urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
urinary tract infection (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
vitrectomy (Eye disorders) | 0 | 0 | 1 | 0 | 0
vitreous degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 1
vitreous detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0
vitreous opacities (Eye disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No